CLINICAL TRIAL: NCT00001727
Title: Screening and Natural History of Patients With Polyostotic Fibrous Dysplasia and the McCune-Albright Syndrome
Status: Recruiting | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980145; 98-D-0145
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01-09

CONDITIONS: McCune-Albright Syndrome
Keywords: Fibrous Dysplasia (FD); McCune-Albright Syndrome (MAS); Natural History
MeSH Terms: conditions — Fibrous Dysplasia, Polyostotic; Fibrous Dysplasia of Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Subjects with Polyostotic Fibrous Dysplasia and McCune-Albright Syndrome.

SUMMARY:
Polyostotic fibrous dysplasia (PFD) is a sporadic disorder which affects multiple sites in the skeleton. The bone at these sites is rapidly resorbed and replaced by abnormal fibrous tissue or mechanically abnormal bone. PFD may occur alone or as part of the McCune-Albright Syndrome (MAS), a syndrome originally defined by the triad of PFD, cafe-au-lait pigmentation of the skin, and precocious puberty. The bony lesions are frequently disfiguring, disabling and painful, and depending on the location of the lesion, can cause significant morbidity. Lesions in weight-bearing bones can lead to disabling fractures, while lesions in the skull can lead to compression of vital structures such as cranial nerves.

The natural history of this disease is poorly described and there are no clearly defined systemic therapies for the bone disease. This is a data collection and specimen acquisition protocol. The purpose of the study is to define the natural history of the disease by following PFD/MAS subjects over time and by using in vitro experimentation with samples/tissue from subjects with the disease.

Study Objectives

1. Primary Objective

   Define the natural history of disease by gaining clinical and basic information about PFD/MAS by following subjects clinically and using in vitro experimentation with tissue from subjects with the disease.
2. Secondary Objective

Refer eligible subjects for enrollment into other appropriate research protocols, if any are currently active.

Study Population

The study population will include:

1. Subjects with known or suspected Polyostotic Fibrous Dysplasia (PFD) or in combination with McCune-Albright Syndrome (MAS)
2. Subjects who meet eligibility criteria will be accepted regardless of gender, race, or ethnicity

Design

This study is an observational/natural history study of PFD/MAS.

Outcome Measures

Primary

1. Successfully enroll subjects with PFD or MAS for the collection, evaluation and analysis of data obtained from clinical visits.
2. Obtain onsite and offsite research tissue (waste tissue) from patients with PFD/MAS that are enrolled onto this study or from individuals with PFD/MAS that are offsite and willing to donate waste tissue to NIH. Research tissue will be used with existing primary cell culture technology (ongoing in our laboratories) to:

   * understand the basic bone biology of the pathologic cell (or cells) involved in the lesions of PFD/MAS
   * determine the presence or absence of mutated cells at "uninvolved sites" to formulate better strategies of predicting the initiation of new lesions, the natural history of lesion progression and/or response to therapy
   * understand osteogenic differentiation, in particular, the role of G(s)alpha in these lesions, which will be transferable to our understanding of bone biology in general
   * understand the pathophysiology of FD and/or endocrine lesions
   * develop better methods of identifying and expanding unaffected bone cells from patients with PFD in an effort to create better grafting material(s)
3. Identify and predict clinical and biological behavior of fibrous dysplastic bone lesions based on:

   * stability, rate of growth, rate of change, progression and regression, and development of new lesions
   * differences between cranial, axial and appendicular lesions
4. Define the natural history of the multiple endocrinopathies associated with MAS and the response to standard of care medications
5. Define clinical and biological aspects of the disease not previously identified
6. Generate future research studies related to PFD alone or in combination with MAS

Secondary

1) Successfully enroll eligible subjects into active research protocols applicable to the FD/MAS population....

DETAILED DESCRIPTION:
Study Description: Polyostotic fibrous dysplasia (PFD) is a sporadic disorder which affects multiple sites in the skeleton. The bone at these sites is rapidly resorbed and replaced by abnormal fibrous tissue or mechanically abnormal bone. PFD may occur alone or as part of the McCune-Albright Syndrome (MAS), a syndrome originally defined by the triad of PFD, cafe-au-lait pigmentation of the skin, and precocious puberty. The bony lesions are frequently disfiguring, disabling and painful, and depending on the location of the lesion, can cause significant morbidity. Lesions in weight-bearing bones can lead to disabling fractures, while lesions in the skull can lead to compression of vital structures such as cranial nerves.

The natural history of this disease is poorly described and there are no clearly defined systemic therapies for the bone disease. This is a data collection and specimen acquisition protocol. The purpose of the study is to define the natural history of the disease by following PFD/MAS subjects over time and by using in vitro experimentation with samples/tissue from subjects with the disease.

Study Objectives

1. Primary Objective

   Define the natural history of disease by gaining clinical and basic information about PFD/MAS by following subjects clinically and using in vitro experimentation with tissue from subjects with the disease.
2. Secondary Objective

Refer eligible subjects for enrollment into other appropriate research protocols, if any are currently active.

ELIGIBILITY:
* INCLUSION CRITERIA

  1. Any patient, age 1 day of life and older, with a likelihood of having PFD or MAS, based on information from an appropriate referring physician or surgeon or provided by the patient or guardian. The diagnosis will be based on typical findings on bone biopsy or on clinical grounds.

EXCLUSION CRITERIA

1. Patient, child, or parent/guardian unwilling to fully cooperate with the evaluations.
2. Patient or parent/guardian unable to provide informed consent.

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with Polyostotic Fibrous Dysplasia and McCune-Albright Syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 1998-12-13 (Actual)

PRIMARY OUTCOMES:
Primary Objective: Define the natural history of disease by gaining clinical and basic information about PFD/MAS by following patients clinically and using in vitro experimentation with tissue from patients with the disease. | 2029
  Successfully enroll, evaluate, and manage subjects with Polyostotic Fibrous Dysplasia and McCune-Albright Syndrome.

SECONDARY OUTCOMES:
Refer eligible patients for enrollment into other appropriate research protocols, if any are currently active. | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Alison M Boyce, M.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Protocol is silent on sharing IPD.

REFERENCES:
- [Derived] Pan KS, FitzGibbon EJ, Vitale S, Lee JS, Collins MT, Boyce AM. Utility of Optical Coherence Tomography in the Diagnosis and Management of Optic Neuropathy in Patients with Fibrous Dysplasia. J Bone Miner Res. 2020 Nov;35(11):2199-2210. doi: 10.1002/jbmr.4129. Epub 2020 Aug 24. PMID 32644197
- [Derived] de Castro LF, Burke AB, Wang HD, Tsai J, Florenzano P, Pan KS, Bhattacharyya N, Boyce AM, Gafni RI, Molinolo AA, Robey PG, Collins MT. Activation of RANK/RANKL/OPG Pathway Is Involved in the Pathophysiology of Fibrous Dysplasia and Associated With Disease Burden. J Bone Miner Res. 2019 Feb;34(2):290-294. doi: 10.1002/jbmr.3602. Epub 2018 Nov 29. PMID 30496606
- [Derived] Robinson C, Estrada A, Zaheer A, Singh VK, Wolfgang CL, Goggins MG, Hruban RH, Wood LD, Noe M, Montgomery EA, Guthrie LC, Lennon AM, Boyce AM, Collins MT. Clinical and Radiographic Gastrointestinal Abnormalities in McCune-Albright Syndrome. J Clin Endocrinol Metab. 2018 Nov 1;103(11):4293-4303. doi: 10.1210/jc.2018-01022. PMID 30124968
- [Derived] Brown RJ, Kelly MH, Collins MT. Cushing syndrome in the McCune-Albright syndrome. J Clin Endocrinol Metab. 2010 Apr;95(4):1508-15. doi: 10.1210/jc.2009-2321. Epub 2010 Feb 15. PMID 20157193
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1998-D-0145.html